CLINICAL TRIAL: NCT05030012
Title: Maintaining Optimal Delivery Using Automatic Titration of Oxygen in Preterm Infants Receiving High Velocity Nasal Insufflation Therapy
Brief Title: Maintaining Optimal HVNI Delivery Using Automatic Titration of Oxygen in Preterm Infants
Acronym: MODERATION Neo
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No path to obtain FDA approval for the legacy Precision Flow OAM.
Sponsor: Vapotherm, Inc. (Industry)
Collaborators: Children's National Research Institute (Other); Seattle Children's Hospital (Other); University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RP-NIOA2019001Reg
Record Dates: First submitted 2021-08-25; First posted 2021-09-01 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Infant, Premature; Neonatal Respiratory Distress; Oxygen Saturation; Bronchopulmonary Dysplasia
Keywords: High Velocity Nasal Insufflation (HVNI); Preterm Infants; Noninvasive Ventilatory Support; Automatic Oxygen Titration; Closed Loop Oxygen Control; High Flow Nasal Cannula
MeSH Terms: conditions — Premature Birth; Pulmonary Atelectasis; Bronchopulmonary Dysplasia | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This study will be a prospective, multi-center, randomized, crossover trial evaluating automated oxygen titration versus manual titration in maintaining oxygen saturation levels in preterm infants requiring noninvasive ventilatory support via high velocity nasal insufflation (HVNI).
Masking Description: This study is unblinded, as there is a distinct difference in modality control between automated and manual modes. Clinical staff are instructed to perform FiO2 adjustments as required, regardless of the study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Automated Control (OAM) (Experimental): In this arm, FiO2 levels delivered via high-velocity nasal insufflation therapy (Vapotherm Precision Flow) will be adjusted by the Oxygen Assist Module (OAM) to keep the infants pulse oxygen saturation within a target range (90-95%). Clinical staff will have the ability to override FiO2 levels when required, and instructed to do so.
  Interventions: Device: Automated Control
- Manual Control (Manual) (Active Comparator): In this arm, FiO2 levels delivered via high-velocity nasal insufflation therapy (Vapotherm Precision Flow) will be manually adjusted by clinical staff to keep infants' oxygen saturation between 90-95%.
  Interventions: Device: Manual Control

INTERVENTIONS:
Device: Automated Control — The purpose of this intervention is to evaluate that the efficacy and safety during the automated performance of the Vapotherm OAM are not inferior to standard care practice (manual control) in maintaining SpO2 levels of 90-95% in preterm infants requiring oxygen adjustments while being treated with high velocity nasal insufflation (HVNI) therapy.
  Other Names: Oxygen Assist Module (OAM); Vapotherm OAM + Vapotherm Precision Flow
  Arms: Automated Control (OAM)
Device: Manual Control — The purpose of this intervention is to establish an active comparator via standard care practice against which to evaluate the efficacy and safety of the automated arm of the study, for determination of non-inferiority of that automated control arm to manual control in maintaining SpO2 levels of 90-95% in preterm infants being treated with high velocity nasal insufflation (HVNI) therapy.
  Other Names: Vapotherm Precision Flow; Treatment as Usual (TAU); Standard of Care (SOC)
  Arms: Manual Control (Manual)

SUMMARY:
Oxygen treatment is common in management of preterm babies requiring intensive care. Delivery of too much or too little oxygen increase the risk of damage to eyes and lungs, and contributes to death and disability. Oxygen control in preterm infants requires frequent adjustments in the amount of oxygen delivered to the baby. This is generally performed manually by a clinician attending the baby, and generally directed to maintaining a specific range of blood oxygen saturation. The manual control often results in only half of the time in the specified range, with the baby experiencing high and low blood oxygen saturations.

The technology being studied is designed to assist the clinician in maintaining blood oxygen saturation within target range by measuring oxygen saturation and automatically adjusting the amount of oxygen delivered for babies receiving high velocity nasal insufflation (an advanced form of high flow oxygen therapy). The proposed study will evaluate the efficacy and safety of the automatic control of oxygen by the new technology, as compared to manual control, among babies receiving high velocity therapy in a neonatal intensive care unit.

DETAILED DESCRIPTION:
Detailed Description: Supplemental oxygen is commonly administered to babies in neonatal intensive care units. The goal of oxygen therapy is to maintain normal oxygenation while minimizing hypoxemia and hypoxemia. Preterm infants are particularly vulnerable to oxygen toxicity and oxidative stress leading to retinopathy of prematurity (ROP), bronchopulmonary dysplasia (BPD), and periventricular leukomalacia (PVL). It's also well known that preterm infants experience hypoxic events exposing the baby to low oxygen levels. These hypoxic events vary as the infant matures, but exposure to prolonged and frequent episodes of hypoxemia is associated with increased morbidity and mortality. The delivery of oxygen is generally controlled by a clinician, and the control decisions are generally made using a non-invasive measure of blood oxygen saturation called pulse oximetry (SpO2) and is a standard of care in the neonatal intensive care unit. The most frequent item adjusted by clinicians to maintain SpO2 within specific target ranges is the fraction of the inspired oxygen (FiO2).

In a recent study by Reynolds, et al., caregiver manual control of oxygen delivered to NICU babies receiving high velocity therapy resulted in only 49% of the total 24-hour study period with the babies within the target SpO2 range (90-95%). by the caregiver based on the monitored oxygen saturation. Similar to the Reynolds findings, Hagadorn et al., conducted a study in 14 centers and showed that preterm infants under 28 weeks' gestation receiving oxygen spent on average only 48% of the time with SpO2 within the prescribed target range, about 36% of the time above and 16% of the time with SpO2 below the target range.

Preterm infants have frequent fluctuations in SpO2 due to their cardio-respiratory instability requiring frequent adjustments of FiO2 . Consequently, these particularly vulnerable infants spend significant time with SpO2 outside the optimal target range and are often exposed to extremes of hypoxemia and hyperoxaemia. The automatic oxygen control system continuously monitors the oxygen saturation and adjusts the oxygen delivery to maintain oxygen saturation within the target range. The efficacy of this mode of oxygen control was demonstrated by Reynolds, et al. in 2018 from two centers in the United Kingdom. Automated control of FiO2 can significantly improve compliance of oxygen saturation targeting and may significantly reduces exposure to hypoxemia as well as hyperoxaemia. The high velocity nasal insufflation therapy is a common mode of non-invasive respiratory support in preterm infants.

Unlike prior studies, this study will include a set of hypothesis-driven safety endpoints (proportion of time above or below target range), stratification by body mass at enrolment, and skin pigmentation phenotype. The objective of this randomized control trial is to evaluate the efficacy of the controller (Vapotherm Oxygen Assist Module [OAM]) in maintaining the SpO2 within target range for premature infants receiving high velocity therapy and presenting with a labile FiO2 requirement.

ELIGIBILITY:
Inclusion Criteria:

1. Infants delivered at a gestational age of less than or equal to 35 6/7 weeks (Preterm) being treated with high velocity nasal insufflation therapy for the management of respiratory distress syndrome
2. Patients that clinically require SpO2 maintenance within the target range of 90-95%
3. A need for supplemental oxygen as demonstrated by a required FiO2 > 0.25 at enrollment
4. Requiring a flow rate of greater than 2 L•min-1 such that the assumed inspired oxygen fraction matched delivered oxygen fraction (definition of HVNI).
5. A minimum of 6 manual FiO2 adjustments in the 24hr period prior to trial enrollment.
6. Willing/Able to complete informed consent.

Exclusion Criteria:

1. Current patient weight of <1000g or >3500g at time of study
2. Major congenital abnormalities
3. Hemodynamic instability, defined as being outside of a normotensive range based on an infant's individual characteristics by clinician
4. Persistent unresolved apnea defined as: requiring 6 stimulations or more per 6 hours
5. Seizures
6. Ongoing sepsis
7. Meningitis
8. Clinician's concern regarding stability of the infant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Billie L Short, MD, Principal Investigator — Children's National Research Institute; Khodayar Rais-Bahrami, MD, Principal Investigator — Children's National Research Institute; Robert J DiGeronimo, MD, Principal Investigator — Seattle Children's Hospital; Robert DiBlasi, RRT-NPS, Principal Investigator — Seattle Children's Hospital; Bradley A Yoder, MD, Principal Investigator — University of Utah Hospital
Locations (3):
- United States (3):
  - Children's National Hospital & Research Institute, Washington D.C., District of Columbia
  - University of Utah Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reynolds PR, Miller TL, Volakis LI, Holland N, Dungan GC, Roehr CC, Ives K. Randomised cross-over study of automated oxygen control for preterm infants receiving nasal high flow. Arch Dis Child Fetal Neonatal Ed. 2019 Jul;104(4):F366-F371. doi: 10.1136/archdischild-2018-315342. Epub 2018 Nov 21. PMID 30464005
- [Background] Hagadorn JI, Furey AM, Nghiem TH, Schmid CH, Phelps DL, Pillers DA, Cole CH; AVIOx Study Group. Achieved versus intended pulse oximeter saturation in infants born less than 28 weeks' gestation: the AVIOx study. Pediatrics. 2006 Oct;118(4):1574-82. doi: 10.1542/peds.2005-0413. PMID 17015549

RESULTS

PARTICIPANT FLOW:
Groups:
- Automated Control (OAM) - Manual Control: The subject started on the Automated Control (OAM) arm. The subject was on this arm for 24 hours. After 24 hours, the subject switched to the Manual Control Arm. The subject was on this arm for 24 hours, for a total of 48 hours.
- Manual Control - Automated Control (OAM): The subject started on the Manual Control arm. The subject was on this arm for 24 hours. After 24 hours, the subject switched to the Automated Control (OAM) arm. The subject was on this arm for 24 hours, for a total of 48 hours.
Period: Overall Study
Arm/Group | Automated Control (OAM) - Manual Control | Manual Control - Automated Control (OAM)
Started | 6 | 9
Completed | 6 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Automated Control (OAM) Then Manual Control: The subjects will start the study on the Automated Control (OAM) for a total of 24 hours. Then, the subjects will switch to the Manual Control Arm for 24 hours, for a total of 48 hours.
- Manual Control (Manual) Then Automated Control (OAM): The subjects will start the study on the Manual Control Arm for a total of 24 hours. Then, the subjects will switch to the Automated Control (OAM) Arm for 24 hours, for a total of 48 hours.
- Total: Total of all reporting groups
Arm/Group | Automated Control (OAM) Then Manual Control | Manual Control (Manual) Then Automated Control (OAM) | Total
Number analyzed (Participants) | 6 | 9 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 9 | 15
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 27.5 (2.8) | 29.7 (3.6) | 28.8 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 2 | 3
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Objective - Percentage of Time Outside of SpO2 Target Range
Description: Percentage of time spent outside target oxygen saturation range, measured by pulse oximetry (SpO2). A lower value indicates a better outcome.
Time Frame: Through study completion, two consecutive 24-hour periods
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Automated Control (OAM) | Manual Control (Manual)
Number analyzed (Participants) | 15 | 15
percentage of time | 24.6 (10.7) | 45.1 (11.4)

2. Primary Outcome: Primary Performance Objective - Percentage of Time Within SpO2 Target Range
Description: Percentage of time spent within target oxygen saturation range, measured by pulse oximetry (SpO2). A higher value indicates a better outcome.
Time Frame: Through study completion, two consecutive 24-hour periods
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Automated Control (OAM) | Manual Control (Manual)
Number analyzed (Participants) | 15 | 15
percentage of time | 73.6 (10.7) | 53.2 (11.8)

3. Secondary Outcome: Performance Endpoint, Percentage of Time IN Range (SpO2 in 90-95% With FiO2 Special at .21) Across the Two Weight Groups.
Description: Percentage of time spent within target oxygen saturation range across two weight groups (1000g-2500g, 2501g-3500g), measured by pulse oximetry (SpO2). A higher value indicates a better outcome.
Time Frame: Through study completion, two consecutive 24-hour periods
Population: There are two weight categories, 14 were in the lower weight and 1 subject was in the higher weight.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Manual Control (Manual) | Automated Control (OAM)
Number analyzed (Participants) | 15 | 15
percentage of time
  Lower Weight (1000g-2500g): number analyzed (Participants) | 14 | 14
  Lower Weight (1000g-2500g) | 52.2 (11.6) | 73.0 (10.9)
  Higher Weight (2501g - 3500g): number analyzed (Participants) | 1 | 1
  Higher Weight (2501g - 3500g) | 67.4 (NA) — There is only one subject in this group - cannot get SD with one data set. | 81.3 (NA) — There is only one subject in this group - cannot get SD with one data set.

4. Secondary Outcome: Secondary Performance Objective 2 - Percentage of Time Within SpO2 Target Range (Skin Pigmentation)
Description: Percentage of time spent within target oxygen saturation range across two skin pigmentation groups (light, dark), measured by pulse oximetry (SpO2). A higher value indicates a better outcome.
Time Frame: Through study completion, two consecutive 24-hour periods
Population: There are two skin pigment groups, dark and light. For the manual arm, there were two subjects in the dark and 13 in the light.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Manual Control (Manual) | Automated Control (OAM)
Number analyzed (Participants) | 15 | 15
percentage of time
  Dark Skin: number analyzed (Participants) | 2 | 2
  Dark Skin | 41.2 (13.8) | 75.7 (19.6)
  Light Skin: number analyzed (Participants) | 13 | 13
  Light Skin | 55.0 (10.9) | 73.3 (10.1)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over the course of the treatment hours, for a total of 48 hours.
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Automated Control (OAM) | Manual Control (Manual)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT05030012/Prot_SAP_000.pdf